CLINICAL TRIAL: NCT01444053
Title: Retrospective Study of the Health Benefits of Ultra-Violet Filtering Contact Lenses
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-201010
Record Dates: First submitted 2011-08-30; First posted 2011-09-30 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Wearers of contact lenses without UV Protection: Subjects who have worn a soft contact lens without UV protection for the past five years or more.
  Interventions: Device: No Intervention
- Wearers of contact lenses with UV Protection: Subjects who have worn a soft contact lens with UV protection for the last 5 years or more.
  Interventions: Device: No Intervention

INTERVENTIONS:
Device: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to examine the long term effect of ultra-violet filtering contact lenses on macular pigment density (MPOD) and accommodative function.

ELIGIBILITY:
Inclusion Criteria:

* The subject is an adapted soft contact lens wearer of at least 5 years duration of either an UV filtering contact lens or a non-UV filtering contact lens
* The subject must report wearing their contact lenses, on average, for a minimum of 5 days each week.
* The subject must have best corrected visual acuity of 6/7.5 or better in each eye.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must read and sign the statement of informed consent
* The subject must be between 18 and 43 years of age

Exclusion Criteria:

* On medication known to affect accommodation
* Active ocular surface pathology
* Had eye surgery
* Significant ocular tissue anomaly
* Any medical condition that may be prejudicial to the study
* Diabetes

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subject selection is based on a history of wearing one of two types of contact lenses for at least five years. Age-matching subjects into 4 age-brackets will be attempted with a target of five subjects in each age bracket among the two types of lenses.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-01 (Actual)

PRIMARY OUTCOMES:
Macular Pigment Optical Density (MPOD) after 5 years of contact lens wear | Approximately 40 minutes
  The MPOD will be assessed at a single visit will be compared between wearers of contact lenses with UV protection and those wearers of lenses without UV protection, based on their 5 year wear history.
Amplitude of Accommodation after 5 years of contact lens wear | Approximately 40 minutes
  Measured with autorefractor at a single visit and will be compared between wearers of contact lenses with UV protection and those wearers of lenses without UV protection, based on their 5 year wear history.

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham, United Kingdom